CLINICAL TRIAL: NCT05633615
Title: A Randomized Phase II Trial of Consolidation Therapy Following CD19 CAR T-Cell Treatment for Relapsed/Refractory Diffuse Large B-Cell Lymphoma or Grade IIIB Follicular Lymphoma
Brief Title: Testing Drug Treatments After CAR T-cell Therapy in Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2114; NCI-2022-07930 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2114 (Other: SWOG); S2114 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Large B-Cell Lymphoma; Grade 3b Follicular Lymphoma; Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Transformed Follic Lymph to Diff Large B-Cell Lymphoma; Transformed Marg Zone Lymph to Diff Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — axicabtagene ciloleucel; Specimen Handling; Cyclophosphamide; fludarabine; Watchful Waiting; Observation; polatuzumab vedotin; Magnetic Resonance Spectroscopy; tisagenlecleucel; CTL019 chimeric antigen receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Step I (lymphodepleting chemotherapy) (Experimental): Patients receive lymphodepleting chemotherapy consisting of fludarabine IV and cyclophosphamide IV on study. Patients then receive tisagenlecleucel IV, axicabtagene ciloleucel IV, or lisocabtagene maraleucel IV on study.
  Interventions: Biological: Axicabtagene Ciloleucel; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Lisocabtagene Maraleucel; Procedure: Positron Emission Tomography; Biological: Tisagenlecleucel
- Step II Arm I (mosunetuzumab) (Experimental): Patients receive mosunetuzumab IV on study. Patients also undergo PET-CT and/or CT and undergo collection of blood and tissue samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Mosunetuzumab; Procedure: Positron Emission Tomography
- Step II Arm II (polatuzumab vedotin) (Experimental): Patients receive polatuzumab vedotin IV on study. Patients also undergo PET-CT and/or CT and undergo collection of blood and tissue samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Polatuzumab Vedotin; Procedure: Positron Emission Tomography
- Step II Arm III (polatuzumab vedotin, mosunetuzumab) (Experimental): Patients receive polatuzumab vedotin IV and mosunetuzumab IV on study. Patients also undergo PET-CT and/or CT and undergo collection of blood and tissue samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Mosunetuzumab; Drug: Polatuzumab Vedotin; Procedure: Positron Emission Tomography
- Step II Arm IV (observation) (Active Comparator): Patients undergo observation on study. Patients also undergo PET-CT and/or CT and undergo collection of blood and tissue samples throughout the study. Patients with subsequent progression within 12 months of CAR T-cell therapy may crossover to Arm III.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Patient Observation; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: Axicabtagene Ciloleucel — Given IV
  Other Names: KTE C19; KTE-C19; KTE-C19 CAR; Yescarta
  Arms: Step I (lymphodepleting chemotherapy)
Procedure: Biospecimen Collection — Undergo collection of blood and tissue samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Step II Arm I (mosunetuzumab); Step II Arm II (polatuzumab vedotin); Step II Arm III (polatuzumab vedotin, mosunetuzumab); Step II Arm IV (observation)
Procedure: Computed Tomography — Undergo PET-CT or CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
  Arms: Step II Arm I (mosunetuzumab); Step II Arm II (polatuzumab vedotin); Step II Arm III (polatuzumab vedotin, mosunetuzumab); Step II Arm IV (observation)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Step I (lymphodepleting chemotherapy)
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
  Arms: Step I (lymphodepleting chemotherapy)
Biological: Lisocabtagene Maraleucel — Given IV
  Other Names: Anti-CD19-CAR Genetically Engineered Autologous T Lymphocytes JCAR017; Anti-CD19-CAR Genetically Engineered Autologous T-lymphocytes JCAR017; Autologous Anti-CD19-EGFRt-4-1BB-zeta-modified CAR CD8+ and CD4+ T-lymphocytes JCAR017; Breyanzi; JCAR 017; JCAR017
  Arms: Step I (lymphodepleting chemotherapy)
Biological: Mosunetuzumab — Given IV
  Other Names: Anti-CD20 x Anti-CD3 Bispecific Monoclonal Antibody BTCT4465A; BTCT 4465A; BTCT-4465A; BTCT4465A; CD20/CD3 BiMAb BTCT4465A; RG 7828; RG-7828; RG7828; RO7030816
  Arms: Step II Arm I (mosunetuzumab); Step II Arm III (polatuzumab vedotin, mosunetuzumab)
Other: Patient Observation — Undergo observation
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
  Arms: Step II Arm IV (observation)
Drug: Polatuzumab Vedotin — Given IV
  Other Names: ADC DCDS4501A; Antibody-Drug Conjugate DCDS4501A; DCDS4501A; FCU 2711; polatuzumab vedotin-piiq; Polivy; RG7596; Ro 5541077-000
  Arms: Step II Arm II (polatuzumab vedotin); Step II Arm III (polatuzumab vedotin, mosunetuzumab)
Procedure: Positron Emission Tomography — Undergo PET-CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Biological: Tisagenlecleucel — Given IV
  Other Names: CART-19; CART19; CTL019; CTL019 T-cells; Kymriah; Tisagenlecleucel-T
  Arms: Step I (lymphodepleting chemotherapy)

SUMMARY:
This phase II trial tests whether mosunetuzumab and/or polatuzumab vedotin helps benefit patients who have received chemotherapy (fludarabine and cyclophosphamide) followed by chimeric antigen receptor (CAR) T-cell therapy (tisagenlecleucel, axicabtagene ciloleucel, or lisocabtagene maraleucel) for diffuse large B-cell lymphoma that has come back (recurrent) or that does not respond to treatment (refractory) or grade IIIb follicular lymphoma. Mosunetuzumab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Polatuzumab vedotin is a monoclonal antibody, called polatuzumab, linked to a drug called vedotin. Polatuzumab is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of cancer cells, and delivers vedotin to kill them. Chemotherapy drugs, such as fludarabine and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. CAR T-cell therapy is a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein on the patient's cancer cells is added to the T cells in the laboratory. The special receptor is called a chimeric antigen receptor. Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. Giving mosunetuzumab and/or polatuzumab vedotin after chemotherapy and CAR T-cell therapy may be more effective at controlling or shrinking the cancer than not giving them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the progression-free survival in participants with relapsed/refractory large B-cell lymphoma or follicular lymphoma grade 3B with stable disease (SD) or partial remission (PR) on first imaging response by central review (day +30 positron emission tomography [PET]/computed tomography [CT] scan) after commercial CD19 CAR T-cell therapy who are randomized to receive each consolidation therapy versus those that receive no consolidation therapy (i.e. control).

Ia. Specifically, to compare the progression free survival (PFS) of 1) mosunetuzumab consolidation to no consolidation, 2) polatuzumab vedotin consolidation to no consolidation, 3) mosunetuzumab + polatuzumab vedotin to no consolidation.

SECONDARY OBJECTIVES:

I. To compare overall survival (OS) in participants randomized to each consolidation treatment arm versus control.

II. To compare the complete remission (CR) conversion rate up to one year in participants randomized to each consolidation arm versus control.

III. To evaluate the treatment-related adverse events in participants randomized to each consolidation arm.

IV. To evaluate the association between total metabolic tumor volume (TMTV), standardized uptake value (SUV) max, and sum product (SPD) of diameters by PET-CT at first imaging response with complete remission conversion up to one year in participants randomized to each consolidation arm as well as those randomized to control.

V. To evaluate the overall response rate (ORR), CR rate, PFS, and OS of participants randomized to Arm 4 (observation) who have lymphoma progression within 12 months of CAR T-cell infusion and subsequently 'cross-over' to receive treatment with mosunetuzumab + polatuzumab vedotin.

VI. To estimate overall survival for all patients registered to this study. VII. To assess the difference in overall survival between participants who achieved CR at first imaging (day +30) versus those who did not achieve CR at first imaging.

BANKING OBJECTIVES:

I. To bank specimens for future correlative studies. II. To bank PET-CT images for future correlative studies.

OUTLINE:

STEP I: Patients receive lymphodepleting chemotherapy consisting of fludarabine intravenously (IV) and cyclophosphamide IV on study. Patients then receive tisagenlecleucel IV, axicabtagene ciloleucel IV, or lisocabtagene maraleucel IV on study.

STEP II: Patients are randomized to 1 of 4 arms.

ARM I: Patients receive mosunetuzumab IV on study. Patients also undergo PET-CT and/or CT and undergo collection of blood and tissue samples throughout the study.

ARM II: Patients receive polatuzumab vedotin IV on study. Patients also undergo PET-CT and/or CT and undergo collection of blood and tissue samples throughout the study.

ARM III: Patients receive polatuzumab vedotin IV and mosunetuzumab IV on study. Patients also undergo PET-CT and/or CT and undergo collection of blood and tissue samples throughout the study.

ARM IV: Patients undergo observation on study. Patients also undergo PET-CT and/or CT and undergo collection of blood and tissue samples throughout the study. Patients with subsequent progression within 12 months of CAR T-cell therapy may crossover to Arm III.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1: REGISTRATION: Participants must have a histologically confirmed diagnosis of diffuse large B-cell lymphoma or follicular lymphoma grade 3b or primary mediastinal large B-cell lymphoma (PMBCL)
* STEP 1: REGISTRATION: Participants with transformed DLBCL must have transformed DLBCL from follicular or marginal zone lymphoma
* STEP 1: REGISTRATION: Participant must have bi-dimensionally measurable systemic disease (at least one lesion with longest diameter > 1.5 cm)
* STEP 1: REGISTRATION: Participants with secondary central nervous system (CNS) lymphoma (parenchymal, spinal cord, meningeal, cerebrospinal fluid involvement) must be asymptomatic from their CNS disease
* STEP 1: REGISTRATION: Participants must be registered for step 1 after they have signed institutional consent for CAR T-cell leukapheresis but prior to the start of lymphodepleting (LD) chemotherapy for commercial CAR T-cell product
* STEP 1: REGISTRATION: In the opinion of the enrolling physician, participants must be felt to be a candidate for CAR T-cell therapy with plans to be treated with Food and Drug Administration (FDA) approved commercially available CD19 CAR T-cell construct.

  * Participants must qualify for commercially approved CD19 CAR T-cell therapy per FDA package insert.
  * If the CAR T-cell product does not meet parameters to be given as an FDA approved product (i.e. does not meet specification criteria mandated by FDA and is infused under an expanded access protocol [EAP] or single participant investigational new drug [IND]) the participant will be taken off of study and no longer be eligible for step 2 randomization
* STEP 1: REGISTRATION: Participants are permitted to receive or have received 'bridging therapy' after CAR T-cell leukapheresis. However, participants must not receive polatuzumab vedotin, and/or mosunetuzumab as part of bridging therapy.

  * Bridging therapy is defined as lymphoma directed therapy administered between leukapheresis and the start of LD chemotherapy. This includes cytotoxic chemotherapy (e.g.: bendamustine and rituximab [BR], rituximab, gemcitabine and oxaliplatin [R-gem/ox]), radiation, corticosteroids, as well as novel therapies such as BTK inhibitors (e.g.: Ibrutinib), immunomodulators (e.g.: lenalidomide), monoclonal antibodies (e.g.: rituximab, obinutuzumab, tafasitamab) antibody drug conjugates (e.g: loncastuximab), checkpoint inhibitors (e.g.: pembrolizumab, nivolumab), clinical trial treatments, etc.
  * If a participant receives polatuzumab vedotin or mosunetuzumab as bridging they will ineligible to continue on step 1 registration portion of the study and be ineligible for step 2 randomization
* STEP 1: REGISTRATION: PET-CT scan must be planned for completion within 60 days prior to the start of LD chemotherapy.

  * All pre-CAR T-cell therapy disease must be assessed and documented on the baseline/pre-registration tumor assessment form.
  * If receiving bridging therapy, participants must have a PET-CT scan upon completion of all planned bridging therapy. If the PET-CT scan after completion of bridging therapy is consistent with complete remission per Lugano criteria as determined by enrolling physician, that participant will be ineligible for step 2 randomization.
  * Participants are permitted to receive corticosteroids after leukapheresis without the need to repeat a PET-CT scan. If steroids are used, they must be planned to stop no later than 3 days before CAR -T cell infusion.
  * If response assessment by central review cannot be completed (I.e., poor quality of PET-CT scan, PET-CT performed out of window, etc.) this would be recorded as 'inadequate assessment' and patient would not be eligible for randomization
* STEP 1: REGISTRATION: Participants that have previously been treated with polatuzumab vedotin or mosunetuzumab prior to CAR T-cell leukapheresis for either indolent or aggressive NHL are eligible as long as the participant did not have refractory disease or progression/relapse within 6 months of the last infusion with either agent
* STEP 1: REGISTRATION: Participants must be planning to receive CAR T-cell infusion no earlier than 2 days and no later than 14 days after completion of the last day of lymphodepleting chemotherapy. Any participant receiving CAR T-cell infusion outside of this window will be ineligible for step 2 randomization
* STEP 1: REGISTRATION: LD chemotherapy prior to CAR T-cell infusion must be planned to start within 60 days after step 1 registration
* STEP 1: REGISTRATION: Participants must be >= 18 years of age at the time of registration
* STEP 1: REGISTRATION: Participants must have Zubrod performance score (PS) of 0, 1, or 2
* STEP 1: REGISTRATION: Total bilirubin =< 2 x institutional upper limit of normal (ULN) (within 14 days prior to registration)

  * Unless due to Gilbert's disease or lymphomatous involvement of liver
* STEP 1: REGISTRATION: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x institutional ULN (within 14 days prior to registration)
* STEP 1: REGISTRATION: Creatinine clearance >= 40 mL/min, as estimated by the Cockcroft and Gault formula. The creatinine value used in the calculation must have been obtained within 14 days prior to registration. Estimated creatinine clearance is based on actual body weight
* STEP 1: REGISTRATION: Participants must have an echocardiogram (ECHO) or multigated acquisition scan (MUGA) within 60 days prior to registration with a cardiac ejection fraction >= 40%.

  * Participants with current symptoms of cardiac disease must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants must be class 2B or better.
  * Participants must not have documented myocardial infarction and percutaneous coronary intervention (PCI) within 6 months prior to registration or myocardial infarction without PCI within 3 months of registration, or unstable angina
* STEP 1: REGISTRATION: Participants with peripheral neuropathy must have < grade 2
* STEP 1: REGISTRATION: Participants with hepatitis B virus infection must have undetectable viral load within 14 days prior to registration, be on suppressive therapy and have no evidence of hepatitis B virus (HBV) related hepatic damage
* STEP 1: REGISTRATION: Participants with hepatitis C infection must have eradication therapy completed, have no evidence of hepatitis C infection (HCV) related damage and have undetectable viral load within 14 days prior to registration
* STEP 1: REGISTRATION: Participants with known human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy at time of registration and have undetectable viral load test on the most recent test results obtained within 6 months prior to registration
* STEP 1: REGISTRATION: Participants must be offered the opportunity to participate in banking for planned translational medicine and future research. With participant consent, any residuals from the mandatory tissue submission will also be banked for future research.

  * Note: Streck tubes must be ordered in advance. Please allow 5-7 days for shipment of the collection kits
* STEP 1: REGISTRATION: NOTE: As a part of the OPEN registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system.

  * Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines.

    * For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations
* STEP 2: RANDOMIZATION: Participants must have met all eligibility criteria for step 1 registration
* STEP 2: RANDOMIZATION: Participant's CAR T-cell product must have met specification parameters to be given as an FDA approved commercial product
* STEP 2: RANDOMIZATION: Participants must have a PET-CT scan between days 25-40 after CAR T-cell infusion and determined to have a response consistent with stable disease or partial remission by central review compared to most recent pre-LD chemo/CAR T-cell PET-CT scan.

  * Note: Patients with delayed enrollment > 21 days after 'day +30' PET-CT scan will necessitate a repeat PET-CT scan if concerning signs or symptoms of lymphoma progression develop.
  * Note: If response assessment by central review cannot be completed (I.e., poor quality of PET-CT scan, PET-CT performed out of window, etc.) this would be recorded as 'inadequate assessment' and patient would not be eligible for randomization
* STEP 2: RANDOMIZATION: Eligible participants must be randomized no later than 60 days after CAR -T infusion
* STEP 2: RANDOMIZATION: Participants must have started LD chemotherapy within 60 days of signing consent for step 1 registration
* STEP 2: RANDOMIZATION: Participants must have S2114 CAR T-cell therapy form submitted to Southwest Oncology Group (SWOG) prior to step 2 randomization
* STEP 2: RANDOMIZATION: Participants must have had a PET-CT scan upon completion of all planned bridging therapy if received, with the exception of up to 7 days of corticosteroids. If the PET-CT scan after completion of bridging therapy was consistent with complete remission per Lugano criteria as determined by enrolling physician, that participant will be ineligible for step 2 randomization.

  * If response assessment by central review cannot be completed (I.e., poor quality of PET-CT scan, PET-CT performed out of window, etc.) this would be recorded as 'inadequate assessment' and patient would not be eligible for randomization
* STEP 2: RANDOMIZATION: Participants must have Zubrod PS of 0, 1, or 2
* STEP 2: RANDOMIZATION: Absolute neutrophil count (ANC) >= 1.0 x 10^3/uL and participants must not have received myeloid growth factor within 72 hours prior to this lab being drawn (within 7 days prior to step 2 randomization)
* STEP 2: RANDOMIZATION: Platelets >= 75 x 10^3/uL and participants must not have received platelet transfusion within 72 hours prior to this lab being drawn (within 7 days prior to step 2 randomization)
* STEP 2: RANDOMIZATION: Total bilirubin =< 2 x institutional ULN (within 7 days prior to step 2 randomization)

  * Unless due to Gilbert's disease or lymphomatous involvement of liver
* STEP 2: RANDOMIZATION: AST and ALT =< 3 x institutional ULN (within 7 days prior to step 2 randomization)
* STEP 2: RANDOMIZATION: Creatinine clearance >= 40 mL/min, as estimated by the Cockcroft and Gault formula. The creatinine value used in the calculation must have been obtained within 7 days prior to step 2 randomization. Estimated creatinine clearance is based on actual body weight (within 7 days prior to step 2 randomization)
* STEP 2: RANDOMIZATION: Participants with peripheral neuropathy must have < grade 2
* STEP 2: RANDOMIZATION: Participants with current symptoms of cardiac disease must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants must be class 2B or better
* STEP 2: RANDOMIZATION: Participants with history of hepatitis B viral infection must have undetectable viral load within 14 days prior to step 2 randomization and on suppressive therapy
* STEP 2: RANDOMIZATION: Participants with history of hepatitis C viral infection must have undetectable viral load within 14 days prior to step 2 randomization
* STEP 2: RANDOMIZATION: Participants with known human immunodeficiency virus (HIV)-infection must be continuing to receive anti-retroviral therapy and have an undetectable viral load test within 14 days prior to step 2 randomization
* STEP 3: CROSSOVER REGISTRATION (ARM 4 ONLY): Participants must have documented disease progression while on Arm 4 (observation) on this protocol. The follow-up tumor assessment form documenting disease progression must be submitted to SWOG prior to step 3 crossover registration
* STEP 3: CROSSOVER REGISTRATION (ARM 4 ONLY): Participants must be registered within 28 days of the date of progression
* STEP 3: CROSSOVER REGISTRATION (ARM 4 ONLY): Participants must have imaging that clearly demonstrates progression compared to day +30 PET-CT scan

  * Note: These scans should be performed as standard of care and only performed between scheduled response assessments required for study if symptoms arise that are concerning for progression
* STEP 3: CROSSOVER REGISTRATION (ARM 4 ONLY): Participants must have Zubrod PS of 0, 1, or 2
* STEP 3: CROSSOVER REGISTRATION (ARM 4 ONLY): ANC >= 1.0 x 10^3/uL and participants must not have received myeloid growth factor within 72 hours prior to this lab being drawn (within 14 days prior to step 3 crossover registration)
* STEP 3: CROSSOVER REGISTRATION (ARM 4 ONLY): Platelets >= 75 x 10^3/uL and participants must not have received platelet transfusion within 72 hours prior to this lab being drawn (within 14 days prior to step 3 crossover registration)
* STEP 3: CROSSOVER REGISTRATION (ARM 4 ONLY): Total bilirubin =< 2 x institutional ULN (within 14 days prior to step 3 crossover registration)

  * Unless due to Gilbert's disease or lymphomatous involvement of liver
* STEP 3: CROSSOVER REGISTRATION (ARM 4 ONLY): AST and ALT =< 3 x institutional ULN
* STEP 3: CROSSOVER REGISTRATION (ARM 4 ONLY): Creatinine clearance >= 40 mL/min, as estimated by the Cockcroft and Gault formula. The creatinine value used in the calculation must have been obtained within days prior to step 3 crossover registration. Estimated creatinine clearance is based on actual body weight (within 14 days prior to step 3 crossover registration)
* STEP 3: CROSSOVER REGISTRATION (ARM 4 ONLY): Participants with peripheral neuropathy must have < grade 2
* STEP 3: CROSSOVER REGISTRATION (ARM 4 ONLY): Participants with current symptoms of cardiac disease must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants must be class 2B or better
* STEP 3: CROSSOVER REGISTRATION (ARM 4 ONLY): Participants with history of hepatitis B viral infection must have undetectable viral load within 14 days prior to step 3 crossover registration and on suppressive therapy
* STEP 3: CROSSOVER REGISTRATION (ARM 4 ONLY): Participants with history of hepatitis C viral infection must have undetectable viral load within 14 days prior to step 3 crossover registration
* STEP 3: CROSSOVER REGISTRATION (ARM 4 ONLY): Participants with known human immunodefici

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From date of randomization to date of first observation of progressive disease or death due to any cause, assessed up to 2 years
  Will compare PFS in participants with relapsed/refractory large B-cell lymphoma or follicular lymphoma grade 3B with stable disease (SD) or partial remission (PR) on first imaging response (day +30 positron emission tomography [PET]/computed tomography [CT] scan) after commercial CD19 chimeric antigen receptor (CAR) T-cell therapy who are randomized to receive each consolidation therapy versus those that receive no consolidation therapy (i.e. control). Specifically, will compare the PFS of 1) mosunetuzumab consolidation to no consolidation, 2) polatuzumab vedotin consolidation to no consolidation, 3) mosunetuzumab + polatuzumab vedotin to no consolidation. Will analyze results by arm rather than assuming no-interactions in some factorial analyses. Will follow multi-step hypothesis testing procedure of Freidlin and Korn to compare the arms within this randomized Phase II study. Each of the primary comparisons has 81% power using a stratified logrank test at one-sided alpha of 0.05.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization to date of death due to any cause, assessed up to 2 years
  Will be estimated using the method of Kaplan-Meier and compared using the stratified log rank test.
Complete remission (CR) conversion rate | Up to 1 year after randomization
  The complete remission conversion rate up to one year after randomization will be calculated and compared using Cochran-Mantel-Haenszel test with a two-sided alpha of .05.
Incidence of adverse events | Up to 2 years
Association between total metabolic tumor volume (TMTV), standardized uptake value (SUV) max, and sum product (SPD) of diameters | Up to 2 years
  The association between TMTV, SUV max, and SPD by PET-CT at first imaging response as a continuous variable will be assessed using a univariate logistic regression with a two-sided alpha of .05, respectively.
Conversion of CR | Up to 2 years
  Evaluated as a binary variable. Assessed using a univariate logistic regression with a two-sided alpha of 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Brian T Hess, Principal Investigator — SWOG Cancer Research Network
Locations (87):
- United States (87):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Highlands Oncology Group - Fayetteville, Fayetteville, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group - Rogers, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UCI Health Laguna Hills, Laguna Hills, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Bronson Battle Creek, Battle Creek, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Case Western Reserve University, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Froedtert and MCW Moorland Reserve Health Center, New Berlin, Wisconsin